CLINICAL TRIAL: NCT03954171
Title: Platino-resistance in Ovarian Cancer
Acronym: PlatinOv
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19 GENF 01
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer; Platinum based-chemotherapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Platinum Compounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with platinum based-chemotherapy (Other)
  Interventions: Other: Patients treated with platinum based-chemotherapy

INTERVENTIONS:
Other: Patients treated with platinum based-chemotherapy — Blood samples, tumor biopsy specimens and ascites samples will be collected at different time points (if feasible, according to the samples taken in the standard practice):
  * before treatment initiation (blood sample),
  * during hospitalisation for surgery (blood sample),
  * during follow-up consultations (blood sample).
  If tumor biopsy and/or ascites sampling are performed during the standard care, a sample will be collected for the study.

SUMMARY:
Prospective, monocentric study aiming to identify factors involved in platinum based-chemotherapy resistance in patients with epithelial ovarian cancer (all stages).

Patients will receive treatment (platinum based-chemotherapy) according to the standard practices.

A prospective database and an associated biological collection will be performed during 5 years:

* For each patient: clinical, biological, epidemiological and therapeutic treatment data will be collected during the standard therapeutic care.
* Biological samples (blood samples, tumor biopsy specimens and ascites samples) will be collected for all patients. These samples will be collected at the same time as those taken in standard practice (no additional biopsy will be performed for the study).

Study participation of each patient will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Epithelial ovarian cancer at initial diagnosis (all stages)
3. Curative treatment (exeresis surgery) not yet initiated excepted neo-adjuvant treatment
4. Indication of platinum based-chemotherapy
5. Patient affiliated to the french social security system
6. Patient must provide written informed consent prior to inclusion in the study and any study-specific procedure

Exclusion Criteria:

1. Non-epithelial ovarian tumor, borderline ovarian tumor
2. Patient with recurrent disease
3. Exploratory surgery not performed at the "Institut Universitaire du Cancer de Toulouse - Oncopole (IUCT-O)"
4. Pregnant or breastfeeding women
5. Any psychological, familial, geographical or sociological condition potentially preventing the medical follow-up and/or study procedures
6. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
The rate of patients alive without progression | 5 years for each patient

SECONDARY OUTCOMES:
The time to onset of platinum based-chemotherapy resistance | 5 years for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France